CLINICAL TRIAL: NCT06357169
Title: Effect of Mechanical Intervention on the Scalp Microbiome: Setting the Stage for the Future Management of Cicatricial Alopecias
Brief Title: Mechanical Intervention on the Scalp Microbiome: Setting the Stage for the Future Management of Cicatricial Alopecias
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: There was only one participant
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: Venus Glow
Record Dates: First submitted 2023-02-27; First posted 2024-04-10 (Actual); Results first posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-01

CONDITIONS: Lichen Planopilaris of Scalp; Alopecia Areata
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Healthy-experimental (Experimental): Healthy participants who have not been diagnosed with scalp or hair disease will be followed over a period of 2 weeks to assess their scalp microbiome and see how well the investigational device works on decreasing the microbe burden of the scalp.
  Interventions: Device: Venus Glow

INTERVENTIONS:
Device: Venus Glow — two treatments over a one week period. At the first visit they will complete an initial questionnaire regarding current scalp care practices, skin type, and hair type. An initial baseline scalp swab and HairMetrix photography in the two swab sites will be taken at the beginning of this visit. Treatment with the Venus Glow™ device will also occur. To treat, the scalp will be divided into four quadrants. Swab samples will be collected at the first baseline and concurrent treatment session, second treatment session and 3-6 days after the last treatment when participants have returned to their usual cleansing routine.

SUMMARY:
The objective of this study is to assess the effect of standardized scalp care, specifically mechanical cleansing with the Venus Glow™ Device and water, on the scalp microbiome. This study also seeks to characterize the microbiome of the normal, healthy scalp, thereby providing a baseline for which the scalp affected by hair and scalp disease can be compared.

DETAILED DESCRIPTION:
The study will assess the effect of mechanical cleansing with the Venus GlowTM Device and water on the scalp microbiome over the course of five in-person visits, each lasting approximately 30-45 minutes. We will test if cleansing the scalp with a mechanical cleansing device changes the composition of the scalp microbiome and improves scalp health. The scalp was swabbed for DNA extraction. Subjects will avoid shampooing, chemical, or heat treatments, but will be able to wet their hair during the study. We also seek to characterize the microbiome of the normal, healthy scalp to provide a baseline for which the scalp affected by hair and scalp disease (e.g., cicatricial alopecia) can be compared.

The first visit will consist of questionnaires about demographics, participants' current hair and scalp practices, skin type, and hair type. The study staff will also swab the mid-frontal regions of the scalp on the right and left sides and take HairMetrix photography. The participant will subsequently undergo Venus GlowTM treatment #1 on the right side of the scalp only. After the treatment, the study staff will re-swab the right side of the scalp. HairMetrix photography in the two swab sites will be taken after each subsequent treatment discussed below.

Visit 2, three days after visit 1, will assess adverse effects, if applicable, from the first treatment. The right side of the scalp will be treated with the Venus GlowTM device again.

Visit 3, three days after visit 2, will also assess adverse effects, if applicable from the second treatment. The study staff will swab the mid-frontal regions of the scalp on the right and left sides. The participant will subsequently undergo Venus GlowTM treatment #3 on the right side of the scalp only. After the treatment, the study staff will re-swab the right side of the scalp.

Visit 4, three days after visit 3, will begin with the adverse effects assessment/check-in. Then, the participant will undergo Venus GlowTM treatment #4 on the right side of the scalp.

Visit 5, approximately two weeks after Visit 1, is the follow-up visit. No treatment will be performed at this last visit. An adverse effects assessment will take place, and the study staff will swab both the right and left mid-frontal regions of the scalp.

ELIGIBILITY:
Inclusion Criteria:

* All individuals between 18-35 years of age
* Ability to understand study procedures and to comply with them

Exclusion Criteria:

* Non-English speakers
* Exclusion related to pregnancy, lactation, or has plans to become pregnant over the course of the study, Based on self-report from the participant
* Current scalp or hair disease diagnosis
* Using oral or topical antimicrobial medication 4 weeks prior to their baseline visit or in the duration of the study
* Current clinical condition that, in the opinion of the site investigator, would interfere with adherence to study requirements
* Inability or unwillingness of individual to give written informed consent

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ronda Farah, MD, Principal Investigator — University of Minnesota; Maria Hordinsky, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Healthy-experimental
Started | 23
Completed | 21
Not Completed | 2

BASELINE CHARACTERISTICS:
Arm/Group | Healthy-experimental
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 23
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.22 (5.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 6
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 14
  More than one race | 2
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Scalp Microbiome Composition
Description: as assessed by relative abundance of genera from scalp swab DNA extraction of the right and left mid-frontal scalp. Kruskal-Wallis will be used to assess variation in microbiome composition between treatment groups
Time Frame: Day 14
Measure: Mean (Standard Deviation); unit: genera
Arm/Group | Healthy-experimental
Number analyzed (Participants) | 21
genera | 10 (0.005)

2. Secondary Outcome: Scalp Health
Description: Blinded scalp health ratings of standardized scalp photos of 15x magnification were completed by two board-certified dermatologists using the Adherent Scalp Flaking Score (0=no scales, 1=thin scales, 2=diffused thin scales, 3=thick heaped-up scales but not forming plaques, 4=diffused thick heaped-up scales but not forming plaques, 5=very thick heaped-up scales forming plaques)
Time Frame: Assessed at day 1 (baseline).
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Healthy-experimental
Number analyzed (Participants) | 21
score | 1.21 (1)

3. Secondary Outcome: Post-treatment 1 Right-sided Scalp Health
Description: as for outcome 2
Time Frame: Assessed at day 7
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Healthy-experimental
Number analyzed (Participants) | 21
score | 1.18 (0.99)

4. Secondary Outcome: Post-treatment 2 Right-sided Scalp Health
Description: as for outcome 2
Time Frame: Assessed at day 14
Measure: Mean (Standard Deviation); unit: score
Arm/Group | Healthy-experimental
Number analyzed (Participants) | 21
score | 1.67 (0.93)

ADVERSE EVENTS:
Time Frame: 2-weeks
Arm/Group | Healthy-experimental
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

LIMITATIONS AND CAVEATS:
The limitations of the trial are as follows: small sample size, short interim between treatment sessions, no scalp/hair disease group.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-05): https://cdn.clinicaltrials.gov/large-docs/69/NCT06357169/Prot_SAP_000.pdf
  • Informed Consent Form (2023-09-29): https://cdn.clinicaltrials.gov/large-docs/69/NCT06357169/ICF_001.pdf